CLINICAL TRIAL: NCT01804946
Title: Multicentre Open Label Comparative Parallel-group Randomized Clinical Trial of Clinical Efficiency and Safety of Ergoferon in Treatment of Influenza
Brief Title: Clinical Trial of Clinical Efficiency and Safety of Ergoferon in Treatment of Influenza
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMH-ER-001
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2013-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — ergoferon; Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ergoferon (1 tablet 3 times a day) (Experimental): 1 tablet per 1 intake: on day 1 of the treatment 8 tablets (1 tablet every 30 minutes for the first 2 hours, then 1 tablet 3 times a day with equal intervals starting on the same day. From day 2 to day 5 1 tablet TID.
  Interventions: Drug: Ergoferon
- Oseltamivir(Tamiflu): 75 mg two times a day. (Active Comparator): Oseltamivir for 5 days (75 mg b.i.d.).
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Ergoferon — Safety and Efficiency of Ergoferon in treatment of Influenza
  Arms: Ergoferon (1 tablet 3 times a day)
Drug: Oseltamivir — Safety and Efficiency in treatment of Influenza
  Other Names: Tamiflu
  Arms: Oseltamivir(Tamiflu): 75 mg two times a day.

SUMMARY:
The purpose of this study is:

* to assess clinical efficiency of Ergoferon for treatment of influenza
* to assess safety of Ergoferon for treatment of influenza
* to compare efficiency of Ergoferon and Tamiflu for treatment of influenza

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged from 18 to 60 inclusively.
2. Patients with body temperature >37,8°C at the moment of examination by the doctor; with at least one catarrh symptom (cough, rhinitis, sore throat) and one intoxication symptom (myalgia, fever/hyperhidrosis, malaise, weakness, headache) during seasonal influenza morbidity.
3. Diagnosed influenza confirmed by express diagnostics (presence of antigens of influenza virus in nasal passages epithelium and proved by QuickVue immunological test).
4. The possibility to start therapy within 24 hours after the onset of the first influenza symptoms.
5. Signed Informed Consent form for participation in the study.

Exclusion Criteria:

1. Patients aged below 18 years and above 60 years.
2. Suspected invasive bacterial infection or presence of severe disease requiring use of antibacterial drugs (including sulfanilamides).
3. Vaccination against influenza prior to epidemic season onset.
4. Medical history of polyvalent allergy.
5. Allergy/ intolerance to any of the components of medications used in the treatment.
6. Exacerbation or decompensation of chronic diseases affecting the patient's ability to participate in the clinical trial.
7. Chronic renal insufficiency.
8. Intake of medicines listed in the section "Prohibited concomitant treatment" for 15 days prior to the inclusion in the trial.
9. Pregnancy, breast feeding, unwillingness to keeping to contraception method during the study.
10. Drug addiction, alcohol usage in the amount over 2 units of alcohol per day.
11. Patients, who from investigator's point o view, will fail to comply with the observation requirements of the trial or with the intake regimen of the investigated medicines.
12. Participation in other clinical trials in the course of 1 month prior to the inclusion in the trial.
13. The patient is related to the research personnel of the investigative site, who are directly involved in the trial or are the immediate relative of the reseacher. The immediate relatives includes husband / wife, parents, children, brothers (or sisters), regardless of whether they are natural or adopted.
14. The patient works for OOO "NPF "Materia Medica Holding" (i.e. is the company's employee, temporary contract worker or designated official responsible for carrying out the research) or the immediate relative.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2011-02; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Putilovskiy, MD, PhD, Study Director — Materia Medica Holding
Locations (8):
- Russia (8):
  - Federal State Budgetary Institution "Scientific Research Institute for Vaccines and Serum named after I.I.Mechnikov" of Russian Academy of Medical Science, Moscow
  - State Budgetary Educational Institution of Higher Professional Education "The Russian National Research Medical University named after N.I. Pirogov" of Ministry of Health and Social Development of Russian Federation, Moscow
  - Federal State Budgetary Institution "Polyclinic № 3" of Affairs Management Department of the President of Russian Federation, Moscow
  - St. Petersburg State Budgetary Health Care Institution "City Polyclinic №106", Saint Petersburg
  - St. Petersburg State Budgetary Health Care Institution "Сity Polyclinic № 117", Saint Petersburg
  - State Budgetary Educational Institution of Higher Professional Education "Smolensk State Medical Academy" of Ministry of Health and Social Development of Russian Federation, Smolensk
  - State Educational Institution of Higher Professional Education "Voronezh State Academy named after N.N. Burdenko" of Ministry of Health and Social Development of Russian Federation, Voronezh
  - State Budgetary Educational Institution of Higher Professional Education "Yaroslavl State Medical Academy" of Ministry of Health and Social Development of Russian Federation, Yaroslavl

REFERENCES:
- [Derived] Rafalsky V, Averyanov A, Bart B, Minina E, Putilovskiy M, Andrianova E, Epstein O. Efficacy and safety of Ergoferon versus oseltamivir in adult outpatients with seasonal influenza virus infection: a multicenter, open-label, randomized trial. Int J Infect Dis. 2016 Oct;51:47-55. doi: 10.1016/j.ijid.2016.09.002. Epub 2016 Sep 8. PMID 27616034

RESULTS

PARTICIPANT FLOW:
Groups:
- Ergoferon Group (EG): Adults aged 18 to 60 years were on the treatment regimen with Ergoferon for 5 days. 1 tablet per 1 intake: on day 1 of the treatment 8 tablets (1 tablet every 30 minutes for the first 2 hours, then 1 tablet 3 times a day with equal intervals starting on the same day. From day 2 to day 5 1 tablet t.i.d.
- Oseltamivir Group (OG): Adults aged 18 to 60 years were on Oseltamivir for 5 days (75 mg b.i.d.).
Period: Overall Study
Arm/Group | Ergoferon Group (EG) | Oseltamivir Group (OG)
Started | 81 | 80
Completed | 79 | 76
Not Completed | 2 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Insufficient data available | 0 | 1
Not completed — Do not meet inclusion criteria | 1 | 2

BASELINE CHARACTERISTICS:
Population: FAS included 78 patients per group: 5 patients excluded with the entry criteria violations (3, EG; 1, OG) and the lack of data (1, OG). PPSet contained 75 patients in EG and 72 ones in OG: 9 were excluded due to protocol violation (3, EG; 2, OG), the failure to satisfy not major entry criteria (3, OG) and due to assigning a prohibited drug (1, OG).
Groups:
- Ergoferon Group (EG): 1 tablet per 1 intake: on day 1 of the treatment 8 tablets (1 tablet every 30 minutes for the first 2 hours, then 1 tablet 3 times a day with equal intervals starting on the same day. From day 2 to day 5 1 tablet TID.
  Ergoferon: Safety and Efficiency of Ergoferon in treatment of Influenza
- Oseltamivir Group (OG): Oseltamivir(Tamiflu): Safety and Efficiency in treatment of Influenza
- Total: Total of all reporting groups
Arm/Group | Ergoferon Group (EG) | Oseltamivir Group (OG) | Total
Number analyzed (Participants) | 81 | 80 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (11.6) | 34.9 (12.6) | 34.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 55 | 104
  Male | 32 | 25 | 57
Region of Enrollment [Number; unit: participants]
  Russian Federation | 81 | 80 | 161

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Normal Body Temperature
Description: Axillary temperature (morning and evening) decline to or below 37.0 ºС (without subsequent increase during ≥24 h)
Time Frame: Day 1 to Day 5
Population: The Per Protocol (PP) set includes subjects received full per protocol therapy, completed all scheduled visits and had no substantial deviations from the protocol. Since PP-analysis and ITT-analysis demonstrated similar (confirmative) results the results of PP-analysis are presented.
Measure: Number; unit: Percentage of participants
Groups:
- Oseltamivir Goup (OG): Oseltamivir(Tamiflu): Safety and Efficiency in treatment of Influenza
Arm/Group | Ergoferon Group (EG) | Oseltamivir Goup (OG)
Number analyzed (Participants) | 75 | 72
Percentage of participants
  Evening, Day 1 | 4 | 1
  Evening, Day 2 | 15 | 15
  Evening, Day 3 | 41 | 43
  Evening, Day 4 | 68 | 72
  Evening, Day 5 | 84 | 88
Statistical Analysis 1: Comparison: Ergoferon Group (EG) vs Oseltamivir Goup (OG); PP set was analyzed; Test type: Non-Inferiority or Equivalence — The pre-determined margin of 20% of the control group effect was used; p = 0.05, Wald method of Z statistics calculation — One-sided, p-value was adjusted for multiple comparisons using the adaptive Holm method; Wald method of Z statistics computed a confidence interval of proportion difference; Risk Difference (RD) = 0

2. Secondary Outcome: Percentage of Patients With Resolution of Influenza Symptoms
Description: Assessment of the proportion of subjects with no clinical symptoms of the disease (fever, common and respiratory symptoms) at Study Day 7 (Visit 3). The severity of influenza symptoms was assessed by a physician with 0 to 3 point scale, where 0 means no symptom, 1=mild symptom, 2=moderate symptom, and 3=severe symptom
Time Frame: on the day 7 of the observation
Population: Per Protocol set.
Measure: Number; unit: Percentage of participants
Groups:
- Ergoferon Group: Adults aged 18 to 60 years were on the treatment regimen with Ergoferon for 5 days. 1 tablet per 1 intake: on day 1 of the treatment 8 tablets (1 tablet every 30 minutes for the first 2 hours, then 1 tablet 3 times a day with equal intervals starting on the same day. From day 2 to day 5 1 tablet t.i.d.
- Oseltamivir Group: Adults aged 18 to 60 years were on Oseltamivir for 5 days (75 mg b.i.d.).
Arm/Group | Ergoferon Group | Oseltamivir Group
Number analyzed (Participants) | 75 | 72
Percentage of participants
  Fever | 100 | 100
  Common symptoms | 61 | 64
  Respiratory symptoms | 83 | 76
  All symptoms | 47 | 49
Statistical Analysis 1: Comparison: Ergoferon Group vs Oseltamivir Group; PP set was analyzed; Test type: Non-Inferiority or Equivalence — The pre-determined margin of 20% of the control group effect was used; p < 0.05, Wald method of Z statistics calculation — One-sided, p-value was adjusted for multiple comparisons using the adaptive Holm method; Wald method of Z statistics computed a confidence interval of proportion difference; Risk Difference (RD) = 0

3. Secondary Outcome: Time to Resolution of the Influenza
Description: Time to resolution was considered as time to the absence of any flu symptom. Absence of symptoms was considered as axillary temperature decline to or below 37.0 ºС without subsequent rise, resolution of the common and respiratory symptoms.
  The duration of a symptom was defined by physician recorded presence/absence of the symptoms during a physical examination at Day 1 to Day 7.
Time Frame: Day 1 to Day 7
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ergoferon Group | Oseltamivir Group
Number analyzed (Participants) | 75 | 72
Days
  Fever | 2.1 (1.4) | 2.3 (1.6)
  Common symptoms | 2.6 (2.2) | 2.4 (2.1)
  Respiratory symptoms | 2.7 (2.5) | 2.6 (2.6)
  All influenza symptoms | 2.6 (2.3) | 2.5 (2.2)
Statistical Analysis 1: Comparison: Ergoferon Group vs Oseltamivir Group; PP set was analyzed; Test type: Non-Inferiority or Equivalence — The clinically significant margin was assumed to be 0.2 of Oseltamivir effect; p < 0.05, t-test, 1 sided — To adjust for multiple comparisons, the adaptive Holm method was used as a way to control type 1 error; Means were compared using the modified two-sample Student t-test including computation of a confidence interval for a difference between means; Mean Difference (Final Values) = 0

4. Secondary Outcome: Mean Body Temperature
Description: The axillary temperature was assessed during a physical examination at Day 1, 3 and 7; axillary temperature was assessed in degrees (Celsius, °С)
Time Frame: on days 1, 3 and 7 of the observation
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Ergoferon Group | Oseltamivir Group
Number analyzed (Participants) | 75 | 72
°C
  Axillary temperature, Day 1 | 38.3 (0.4) | 38.3 (0.4)
  Axillary temperature, Day 3 | 37.0 (0.5) | 37.0 (0.5)
  Axillary temperature, Day 7 | 36.5 (0.2) | 36.6 (0.3)
Statistical Analysis 1: Comparison: Ergoferon Group vs Oseltamivir Group; PP set was analyzed; Test type: Non-Inferiority or Equivalence — The clinically significant margin was assumed to be 0.2°C; p < 0.05, t-test, 1 sided — To adjust for multiple comparisons, the adaptive Holm method was used as a way to control type 1 error; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0, Standard Deviation 0.5

5. Secondary Outcome: Severity of Influenza Symptoms (Total Score of the Common Symptoms and Respiratory Symptoms)
Description: The severity of influenza symptoms was assessed during a physical examination at Day 1, 3 and 7; common (10 symptoms) and respiratory (5 symptoms) symptom's total score was assessed with using the point scale: 0=No symptom; 1=Mild symptom; 2=Moderate symptom ; 3=Severe symptom. The Common Symptoms total score ranged from 0 (no symptoms) to 30 (severe symptoms). The Respiration Symptoms total score ranged from 0 (no symptoms) to 15 (severe symptoms)
Time Frame: on days 1, 3 and 7 of the observation
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ergoferon Group | Oseltamivir Group
Number analyzed (Participants) | 75 | 72
Scores on a scale
  Common symptoms, Day 1 | 19.0 (6.7) | 18.6 (6.3)
  Common symptoms, Day 3 | 9.2 (5.1) | 7.8 (4.3)
  Common symptoms, Day 7 | 2.3 (2.7) | 1.9 (2.3)
  Respiratory symptoms, Day 1 | 6.1 (3.7) | 5.9 (3.6)
  Respiratory symptoms, Day 3 | 4.3 (2.4) | 4.0 (2.7)
  Respiratory symptoms, Day 7 | 1.3 (1.5) | 1.4 (1.8)
Statistical Analysis 1: Comparison: Ergoferon Group vs Oseltamivir Group; PP set was analyzed; Test type: Non-Inferiority or Equivalence — The margin of no clinical importance was assumed to be 0.5 point or less to assess any symptom based on 4 point scale; p < 0.05, t-test, 1 sided — To adjust for multiple comparisons the adaptive Holm method was used as a way to control type 1 error; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0

6. Secondary Outcome: The Number of the Antipyretic Intake
Description: A subject recorded the number of antipyretic intake in patient diary.
Time Frame: Day 1 to Day 5
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: Number of Doses
Arm/Group | Ergoferon Group | Oseltamivir Group
Number analyzed (Participants) | 75 | 72
Number of Doses
  Day 1 | 0.65 (0.48) | 0.72 (0.45)
  Day 2 | 0.40 (0.49) | 0.49 (0.50)
  Day 3 | 0.19 (0.39) | 0.15 (0.36)
  Day 4 | 0.01 (0.12) | 0.03 (0.17)
  Day 5 | 0.00 (0.00) | 0.01 (0.12)
Statistical Analysis 1: Comparison: Ergoferon Group vs Oseltamivir Group; PP set was analyzed; Test type: Non-Inferiority or Equivalence — To compare the number of antipyretic intake the margin of no clinical importance was assumed to be 0.2; p < 0.05, t-test, 1 sided — To adjust for multiple comparisons, the adaptive Holm method was used as a way to control type 1 error; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0, Standard Deviation 0.5

7. Secondary Outcome: Change in the Patient's Quality of Life.
Description: The quality of life was assessed in influenza patients at baseline and at the end of the treatment period using the European Quality of Life Questionnaire (EQ5D) measuring the health status by five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression (each dimension is assessed by 1 to 3 point scale; the minimum score 5 points refers to the best status, 15 points refers to the worst status).
Time Frame: Day 7 vs. Day 1
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ergoferon Group | Oseltamivir Group
Number analyzed (Participants) | 75 | 72
Scores on a scale
  Day 1 | 9.5 (1.9) | 9.4 (2.2)
  Day 7 | 5.4 (0.9) | 5.4 (0.8)
Statistical Analysis 1: Comparison: Ergoferon Group vs Oseltamivir Group; PP set was analyzed; Test type: Non-Inferiority or Equivalence — To compare the quality of life total score the margin of no clinical importance was assumed to be 0.2 of Oseltamivir group value; p < 0.05, t-test, 1 sided — To adjust for multiple comparisons, the adaptive Holm method was used as a way to control type 1 error; The changes of means (Day 7 vs Day 1) were compared using the modified two-sample Student t-test including computation of a confidence interval; Mean Difference (Final Values) = 0, Standard Deviation 2.2

8. Secondary Outcome: Change in the Subjective Health Status
Description: The patient subjective health status assessment was based on Visual Analogue Scale - VAS). VAS includes a rating of current health status from 0 (worst) to 100 (best).
Time Frame: Day 7 vs. Day 1
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ergoferon Group | Oseltamivir Group
Number analyzed (Participants) | 75 | 72
Scores on a scale
  Day 1 | 41.6 (18.2) | 46.2 (15.4)
  Day 7 | 87.7 (10.7) | 88.0 (10.6)
Statistical Analysis 1: Comparison: Ergoferon Group vs Oseltamivir Group; PP set was analyzed; Test type: Non-Inferiority or Equivalence — To compare the patient subjective health status assessment the margin of no clinical importance was assumed to be 0.2 of Oseltamivir group value; p < 0.05, t-test, 1 sided — To adjust for multiple comparisons, the adaptive Holm method was used as a way to control type 1 error; Changes of means (Day 7 vs Day 1) were compared using the modified two-sample Student t-test including computation of a confidence interval; Mean Difference (Final Values) = 0, Standard Deviation 18.2

9. Secondary Outcome: Percentage of Patients With Complications of the Influenza
Description: Pneumonia, sinusitis, otitis media are examples of the influenza complications
Time Frame: Day 1 to Day 7
Population: Per Protocol set
Measure: Number; unit: Percentage of participants
Arm/Group | Ergoferon Group | Oseltamivir Group
Number analyzed (Participants) | 75 | 72
Percentage of participants | 0 | 2
Statistical Analysis 1: Comparison: Ergoferon Group vs Oseltamivir Group; PP set was analyzed; Test type: Non-Inferiority or Equivalence — The clinically significant difference (margin) between two percentages was assumed to be 20% or more of the effect of Oseltamivir; p < 0.05, The Wald method of Z statistics calcul; The Wald method of Z statistics calculation was performed including computation a confidence interval for a difference between proportions; Risk Difference (RD) = 0

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were registered from Day 1 to Day 7 and during 30 days after the end of the research
Description: Adverse/Serious adverse events were registered in patients of the Full Analysis Set (n=161, Safety Population)
Arm/Group | Ergoferon Group | Oseltamivir Group
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/80
Other Adverse Events (participants affected / at risk) | 11/81 | 15/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergoferon Group (N=81) | Oseltamivir Group (N=80)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Throat burning sensation of (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abnormal feces (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Monocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Urine mucous (Renal and urinary disorders) | 3 (3) | 1 (1)
Proteinuria (Renal and urinary disorders) | 4 (4) | 4 (4)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine white blood cells increased (Investigations) | 2 (2) | 1 (1)
Urine red blood cells increased (Investigations) | 2 (2) | 2 (2)
Crystal urine (Investigations) | 1 (1) | 0 (0)
Bacteria urine (Investigations) | 2 (2) | 1 (1)
Specific gravity urine increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
Bilirubin increased (Investigations) | 2 (2) | 0 (0)
Blood monocytes increased (Investigations) | 1 (1) | 0 (0)
ESR increased (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other